CLINICAL TRIAL: NCT04220099
Title: Pretreatment Electroencephalogram (EEG) May Predict Electroconvulsive Therapy(ECT) Effect in Schizophrenia
Brief Title: Electroencephalogram (EEG) and Electroconvulsive Therapy(ECT) Response in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Other Study IDs: SMHC-SZD-001
Record Dates: First submitted 2019-12-30; First posted 2020-01-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- schizophrenia patients needed ECT treatment: Whether patients need ECT treatment are assessed by clinicians according to American Psychiatric Association(APA) guidelines.
  Interventions: Procedure: Electroconvulsive therapy(ECT)

INTERVENTIONS:
Procedure: Electroconvulsive therapy(ECT) — Patients recieve 8-sessions ECT treatments and those kinds of drugs they take since they were recruited remain unchanged during this study.

SUMMARY:
This study is designed to find quantitative Electroencephalogram(qEEG) biomarkers to predict Electroconvulsive Therapy(ECT) Response in Schizophrenia

DETAILED DESCRIPTION:
The purpose of this proposal is to explore quantitative Electroencephalogram(qEEG) biomarkers that would predict Electroconvulsive Therapy(ECT) Response in Schizophrenia (SZD). The investigators will recruit 30 SZD patients who are preparing for ECT treatment and assesse psychotic symptoms using Positive and Negative symptom scale(PANSS) before and after 8-sessions clinical course of ECT treatment. These patients needed ECT treatment are assessed by clinicians according to American Psychiatric Association(APA) guidelines. Meanwhile resting EEG will be recorded for 10 minutes before the first episode of ECT treatment. Decrease of PANSS scores will be calculated after the last session of ECT treatment to distinguish responder/non-responder.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 criteria for SZD
* patients needed ECT treatment assessed by clinicians using American psychological Association(APA) guidelines.
* symptoms must be of at least moderate severity (PANSS score >71)
* age between 18 to 60 years old
* medications will be stable for at least four weeks prior to ECT, and there will be no dose changes unless medically necessary

Exclusion Criteria:

* any additional current psychiatric comorbidity
* pregnancy or prepare to have a baby
* current use of any Antiepileptic drugs
* history of taking any kinds of Physicotherapeutics within 6 months
* severe psychotic symptoms that make patients could not accomplish the clinical interview

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: schizophrenia patients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-07-04 (Actual)

PRIMARY OUTCOMES:
Change in Positive and negative syndrome scale（PANSS）score | up to 4 weeks
  It assessed the severity of psychotic symptoms.The responder on PANSS is defined as a PANSS decrease at least 25% from the baseline at post-treatment. PANSS helps us divide cases into response and nonresponse group.
EEG functional connectivity difference between response and nonresponse group | through study completion, an average of 6 months
  This is a predictive indicator collected before ECT treatment. After treatment, we divided 30 patients into response and nonresponse group using PANSS. Then we explore differences in pretreatment EEG functional connectivity at different frequency bands (Alpha, Beta, Delta, and Theta) to find a predictable biomarker for ECT treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, Ph.D M.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China